CLINICAL TRIAL: NCT02618694
Title: Posterior Retroperitoneoscopic Approach Versus Transperitoneal Laparoscopic Approach in Management of Adrenal Tumors: A Randomized Comparative Study
Brief Title: Efficacy and Safety of Posterior Retroperitoneoscopic Adrenalectomy: A Comparative Study
Acronym: PostLapAdrnl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Bakr Arabi, Demonstrator, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2380
Record Dates: First submitted 2015-11-15; First posted 2015-12-01 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Adrenal Mass; Adrenal Disease; Pheochromocytoma; Cushing Syndrome
Keywords: adrenal; supra-renal; adrenalectomy; retroperitoneoscopy; posterior retroperitoneoscopy; Laparoscopic adrenalectomy
MeSH Terms: conditions — Adrenal Gland Diseases; Pheochromocytoma; Cushing Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): patient had posterior retroperitoneoscopic adrenalectomy
  Interventions: Procedure: Posterior retroperitoneoscopic adrenalectomy
- Group 2 (Active Comparator): patient had Transperitoneal laparoscopic adrenalectomy
  Interventions: Procedure: Transperitoneal laparoscopic adrenalectomy

INTERVENTIONS:
Procedure: Posterior retroperitoneoscopic adrenalectomy — Patient is in prone, half Jack-knife position, and hips and knees are fixed in 75-90°. A 15 mm trocar incision just below the tip 12th rib. Prepare a small retroperitoneal space with finger and insert two 5 mm trocars about 5 cm lateral and medial to the first trocar with digital guidance. Medial trocar will be inserted upward. Lateral one will be lateral and below the 11th rib. Dissect inferior to diaphragm and retraction of the kidney downward. Mobilize the adrenal gland. At right side, start medial and caudally. Control the adrenl arteries crossing the IVC posteriorly. Prepare adrenal vein posterolaterally. Control between two clips. Continue gland dissection laterally and cranially. At left side, prepare the adrenal vein between the gland and diaphragm medial to the upper pole of the kidney. Dissect medial, lateral and cranially. Retrieve the mass through middle incision. Insert a drain and close skin incisions (Walz M. K., 2005).
  Other Names: Posterior retroperitoneal laparoscopic adrenalectomy
  Arms: Group 1
Procedure: Transperitoneal laparoscopic adrenalectomy — On right side, patient is on supine position. Put a trocar at umbilicus for the camera. Put 4 trocars 1-2 cm subcostal from subxiphoid (10-12 mm) for liver retractor, to far lateral (5 mm) and two 10 mm trocars inbetween. Retract liver, incise the retroperitoneum, and identify right adrenal gland between upper pole of the kidney and IVC. Dissect gland from the kidney than laterally and posteriorly from the diaphragm. Expose, apply clips to, and divide the adrenal vein. On left side, patient is on lateral decubitus. Put a trocar at umbilicus for the camera, 4 trocars 1-2 cm subcostal from the midline to the far most lateral possible (the last is 5 mm the rest are 10 mm). Mobilize colon flexure and expose the kidney. Separate kidney from the pancreas and spleen. Mobilize the tumor, starting by posterior surface, superior border then from the renal surface. Divide the adrenal vein. Retrieve the mass (Suzuki, Tsuru, & Ihara, 2012; Linos, 2005; George & Kavoussi, 2010).
  Other Names: Anterior laparoscopic adrenalectomy; Lateral laparoscopic adrenalectomy
  Arms: Group 2

SUMMARY:
This randomized comparative study assesses the safety and efficacy of the posterior retroperitoneoscopic adrenalectomy in comparison to the standard, anterior transperitoneal approach and suppose that this new technique is a safe and effective alternative to the standard approach.

DETAILED DESCRIPTION:
Aim of the study:

To upgrade the urosurgical care level for candidate of surgical adrenalectomy due to adrenal diseases, to increase efficacy of the procedure and shorten the operative time and duration of hospital stay and convalescence.

Study Objective:

Comparing the safety and efficacy of posterior retroperitoneoscopic versus anterior transperitoneal adrenalectomy, as regard to the operative time, estimated intraoperative blood loss, days of postoperative hospital stay, and rate of complications.

Study Question:

Can the posterior retroperitoneoscopic approach provide a better alternative to anterior laparoscopic approach in terms of effectiveness and safety for laparoscopic adrenalectomy?

Study Hypothesis:

Investigators suggest that posterior retroperitoneoscopic approach is a safe and effective alternative to anterior transperitoneal approach for adrenalectomy with less operative time, estimated blood loss, postoperative days of hospitalization and rate of complications.

Significance and Relevance:

This study is suspected to be beneficial for urologists and oncology surgeons, as they can select the most effective intervention for patients with adrenal disease.

Study setting:

The study will be carried out over one year starting from 4/2015 to 5/2016, including the operations and data management. Operative procedures will be carried out at Urology Departments on Suez Canal, and Alexandria University hospitals.

Study population The study will focus on patients with adrenal disease indicated for adrenalectomy. The sample frame will include patients of any age, gender and body weight, with fair cognitive function, who is candidate for simple laparoscopic adrenalectomy in Suez Canal University Hospital and Alexandria University Hospital. Inclusion and exclusion criteria will be mentioned at Eligibility section.

Sampling:

A non-probability convenience sample will be taken. That is the cases present and referred to urology clinic and diagnosed to have adrenal mass or hyperplasia and are candidates for laparoscopic adrenalectomy.

The sample size will be calculated to compare mean values of two independent groups of equal sizes with a possibility of two way outcome. The sample size will be 20 cases, randomly divided into 10 cases for each group.

Work plan:

The main objective of the study is to compare the data related obtained in the two laparoscopic approachs in order to assess the efficacy of each one and determine a statistic evidence of preferring one of them over the other. This goal could be achieved through the following steps. First, patient evaluation; and this will be through the urology clinic of the university hospitals in Suez Canal and Alexandria Universities. It also includes patients referred from related clinics of oncosurgery, gynecology, endocrinology and cardiology clinics. History taking, full clinical examination will be done. Laboratory investigations will be requested according to provisional clinical diagnosis. Imaging studies will be done to confirm final diagnosis and determine the treatment plan. Second, as the case is indicated and fit for laparoscopic adrenalectomy, and as the case fulfill the inclusion criteria of the study, the patient will get a study number and will be randomly assigned to each operative approach. Third phase of the study is postoperative follow up. The patient will be followed for a month. Parameters will include the postoperative days to full diet, days to mobilization, days to discharge and days to full recovery. Also the postoperative pain score and the scar cosmetic outcome are included.

Instruments:

The theatre room should be prepared for laparoscopic procedure with: a charge-coupled device video camera, a video monitor, Xenon light source, high frequency generator and suction and irrigation devices. Laparoscopic surgeries depend on five main steps. Insufflation using CO2 high flow insufflator. This step involve 2 techniques; the closed techniques with Veress needle in transperitoneal access; and the open Hasson techniques. Trocar insertion that include the multiport type, open or closed technique, retroperitoneal and transperitoneal. Dissection through abdominal planes will need endoscopic curved scissors with or without rotatable blades, endoscopic curved dissectors and suction irrigation probe. Also the procedure may include sharp dissection with endoshears or blunt dissection with endo-peanuts, right angle dissector. Upon heamostasis the basic instruments are: 5 mm monopolar coagulation forceps/dissector, 5 mm bipolar forceps, 10 mm endoclip applicator and endoscopic staplers. LigaSure™ for blunt dissection and heamostasis. Endoscopic needle holder and short threaded small needle are needed for suturing. Finally, the LapSac™ is the best tested bag for retrieval of specimens. The data of the patient and his preoperative and postoperative parameters will be collected by a questionnaire designed for the purposes of this study. It also include the traditional numerical rating scale and visual analogue scale for assessment of the postoperative pain. The patient satisfaction of the scar will be assessed by three questionnaires; body image questionnaire, photo series questionnaire and future surgical procedure preference questionnaire.

Variables:

For each case the data will include demographic data of the patient and his medical and surgical history. This includes age, gender, body mass index calculated as kg/square meter. The side of the affected gland plays a role in operative time, so determination of the side by computed tomography (CT) is essential. Also size of the adrenal mass in CT and the clinical diagnosis regarding the function and the possibility of malignancy will also be considered the main independent variable. A significant independent variable is the surgeon's experience. The number and type of the procedures done by the operator with rate and cause of conversions will be included to each case. Dependent variables will include the full operative data of each case. Starting from the indication of the intervention and the rationale for preference of laparoscopic approach and eventually the cause of conversion if needed. This study focuses on operative time in minutes; total time from the first abdominal incision to the last suture, and the time elapsed to identify the adrenal vein, a critical step at the operation. The study is also interested in comparing the estimated blood loss measured in milliliters and the correlation to the type of tumor, patients and operative variables. On the postoperative phase, the data gathered include the number of days to full diet, of post-operative hospital stay and to complete recovery; i.e. return to usual daily activity. The patient will achieve a score assessment of the postoperative pain and assessment of cosmotic outcome of the incisions. The rate of short term complications postoperatively will be assessed for each group and classified by Clavien-Dindo system.

Statistical Analysis:

This will include data management and coding. The data entry will be via SPSS™ or Microsoft™ Excel™. Mainly the comparison of the study variables will be via detecting the significance of differences between mean values of each group parameters. Finally, the data will be arranged into tables and graphs and presented to conclude the findings of the study.

Ethical consideration:

All patients are informed about participation in training course for urology trainees as a part of the consent of admission and getting surgical intervention at an authorized teaching hospital. However, each participant will be offered an informed consent for being included into this comparative study. The patient will receive his ideal and best line of treatment according to the latest guidelines and available facilities whatever his response to the consent. The risk of complications of both intervention is comparable and all participants will have the same chance to have either transperitoneal or posterior retroperitoneal approaches. To avoid bias, patient will be assigned randomly into the two study groups. At the other hand, patient's data involved at this study will be treated confidentially.

Budget:

This study is funded by the researcher's financial resources. That includes transportation fees, paper work and audio-video utilities. Cases done in the Suez Canal University Hospital may be afforded by the college or the hospital fund. This includes the admission, the rent of the laparoscopic set and the associated medications.

ELIGIBILITY:
Inclusion Criteria: patients have one or more of the following;

* Functioning adrenal adenoma,
* Nonfunctioning adenoma < 7 cm by pelvi-abdominal CT,
* Secondary metastatic adrenal mass suitable for laparoscopic adrenalectomy,
* Adrenal hyperplasia indicated for laparoscopic adrenalectomy.

Exclusion Criteria:

* Patients with cardiovascular disease (as angina, acute myocardial infection, congestive heart failure); history of stroke, transient myocardial attacks, coronary angioplasty or coronary artery bypass graft surgery, or any other contraindication for laparoscopy e.g. COPD,
* Pregnant females,
* Locally advanced malignant disease,
* Evidence of regional lymph node involvement,
* Vascular malignant invasion,
* Malignant uncontrolled hypertension with pheochromocytoma,
* Need for other simultaneous surgical intervention at the same session e.g. cholecystectomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mean operative time | 1 year
  total time from the first abdominal incision to the last suture, and the time elapsed to identify the adrenal vein, a critical step at the operation.
Mean amount of intraoperative blood loss | 1 year
  measured in milliliters.
Mean days of postoperative hospital stay | 1 year
  include the number of days to full diet, to mobilization and to complete recovery; i.e. return to usual daily activity.
Rate of complications | 1.5 year
  classified by Clavien-Dindo classification system

SECONDARY OUTCOMES:
Mean of postoperative pain score | 1 year
  using visual analogue scale or face scale score (according to participant's level of education)
mean of scar cosmetic assessment score | 1.1 year
  The patient satisfaction of the scar will be assessed by THE SUM of scores of three questionnaires; body image questionnaire score + photo series questionnaire score + future surgical procedure preference questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Sami M Shaaban, Professor, Study Chair — Suez Canal University - Department of Urology and Andrology; Haitham M Badawy, PhD, Study Director — Alexandria University - Department of Urology; Tamer H Abou-Youssif, PhD, Study Director — Alexandria University - Department of Urology
Locations (2):
- Egypt (2):
  - Alexandria Main University Hospital, Alexandria, Alexandria Governorate
  - Suez Canal University Hospital, Ismailia, Ismailia Governorate

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Constantinides VA, Christakis I, Touska P, Palazzo FF. Systematic review and meta-analysis of retroperitoneoscopic versus laparoscopic adrenalectomy. Br J Surg. 2012 Dec;99(12):1639-48. doi: 10.1002/bjs.8921. Epub 2012 Sep 28. PMID 23023976
- [Background] Dickson PV, Alex GC, Grubbs EG, Ayala-Ramirez M, Jimenez C, Evans DB, Lee JE, Perrier ND. Posterior retroperitoneoscopic adrenalectomy is a safe and effective alternative to transabdominal laparoscopic adrenalectomy for pheochromocytoma. Surgery. 2011 Sep;150(3):452-8. doi: 10.1016/j.surg.2011.07.004. PMID 21878230
- [Background] Dickson PV, Jimenez C, Chisholm GB, Kennamer DL, Ng C, Grubbs EG, Evans DB, Lee JE, Perrier ND. Posterior retroperitoneoscopic adrenalectomy: a contemporary American experience. J Am Coll Surg. 2011 Apr;212(4):659-65; discussion 665-7. doi: 10.1016/j.jamcollsurg.2010.12.023. PMID 21463807
- [Background] Doublet, J. D., Janetscek, G., Joyce, A., Mandressi, A., Rassweiller, J., & Tolley, D. (2002). Guidelines in laparoscopy. European Association of Urology.
- [Background] Eichel, L., & Clayman, R. V. (2012). Fundamentals of laparoscopic and robotic urologic surgery. In A. J. Wein, S. R. Kavoussi, A. C. Novick, A. W. Partin, & C. A. Peters, Campell and Walsh Urology (pp. 204-253). Philadelphia: Saunders.
- [Background] Ekstein P, Szold A, Sagie B, Werbin N, Klausner JM, Weinbroum AA. Laparoscopic surgery may be associated with severe pain and high analgesia requirements in the immediate postoperative period. Ann Surg. 2006 Jan;243(1):41-6. doi: 10.1097/01.sla.0000193806.81428.6f. PMID 16371735
- [Background] George, A. K., & Kavoussi, L. R. (2010). Laparoscopic Adrenalectomy. In S. D. Graham, T. E. Keane, S. D. Graham, & T. E. Keane (Eds.), Glenn's Urologic Surgery (pp. 859-866). Phiadelphia: Lippincott Williams and Wilkins.
- [Background] Linos, D. (2005). Left anterior laparoscopic adrenalectomy. In D. Linos, & J. A. van Heerden, Adrenal Glnads (pp. 320-324). Berlin: Springers.
- [Background] Linos, D. (2005). Right anterior laparoscopic adrenalectomy. In D. Linos, & J. A. van Heerden, Adrenal Galnd (pp. 313-319). Berlin: Springer.
- [Background] Linos, D., & van Heerden, J. A. (2005). Adrenal Glands: diagnostic aspects and surgical therapy. Berlin: Springer.
- [Background] Manabe D, Saika T, Ebara S, Uehara S, Nagai A, Fujita R, Irie S, Yamada D, Tsushima T, Nasu Y, Kumon H; Okayama Urological Research Group, Okayama, Japan. Comparative study of oncologic outcome of laparoscopic nephroureterectomy and standard nephroureterectomy for upper urinary tract transitional cell carcinoma. Urology. 2007 Mar;69(3):457-61. doi: 10.1016/j.urology.2006.11.005. PMID 17382144
- [Background] Naya Y, Nagata M, Ichikawa T, Amakasu M, Omura M, Nishikawa T, Yamaguchi K, Ito H. Laparoscopic adrenalectomy: comparison of transperitoneal and retroperitoneal approaches. BJU Int. 2002 Aug;90(3):199-204. doi: 10.1046/j.1464-410x.2002.02845.x. PMID 12133053
- [Background] Park SK, Olweny EO, Best SL, Tracy CR, Mir SA, Cadeddu JA. Patient-reported body image and cosmesis outcomes following kidney surgery: comparison of laparoendoscopic single-site, laparoscopic, and open surgery. Eur Urol. 2011 Nov;60(5):1097-104. doi: 10.1016/j.eururo.2011.08.007. Epub 2011 Aug 12. PMID 21856076
- [Background] Sam, A., & Meeran, K. (2009). Licture notes: Endocrinology and Diabetes. UK: Wiley-Black Well.
- [Background] Shalhav AL, Dunn MD, Portis AJ, Elbahnasy AM, McDougall EM, Clayman RV. Laparoscopic nephroureterectomy for upper tract transitional cell cancer: the Washington University experience. J Urol. 2000 Apr;163(4):1100-4. PMID 10737474
- [Background] Suzuki, K., Tsuru, N., & Ihara, H. (2012). Laparoscopic approaches for Adrenal galnds. In J. A. Smith, S. S. Howards, & G. M. Preminger, Hinman's Atlas of Urologic Surgery (pp. 1111-1122). Philadilphia: Sunders.
- [Background] Walz, M. K. (2005). Posterior retroperitoneoscopic adrenalectomy. In D. Linios, & J. A. van Heerden, Adrenal Glands (pp. 333-339). Berlin: Springer.
- [Background] Walz MK, Alesina PF, Wenger FA, Deligiannis A, Szuczik E, Petersenn S, Ommer A, Groeben H, Peitgen K, Janssen OE, Philipp T, Neumann HP, Schmid KW, Mann K. Posterior retroperitoneoscopic adrenalectomy--results of 560 procedures in 520 patients. Surgery. 2006 Dec;140(6):943-8; discussion 948-50. doi: 10.1016/j.surg.2006.07.039. PMID 17188142